CLINICAL TRIAL: NCT05999227
Title: 68Ga-FAPI-04 PET Imaging in Early Response Evaluation of Rectal Cancer Patients Treated With Immunotherapy: A Single-center Clinical Study
Brief Title: 68Ga-FAPI-04 PET Imaging in Early Response Evaluation of Rectal Cancer Patients Treated With Immunotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XLan-0379
Record Dates: First submitted 2023-07-19; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-06

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — 68Ga-FAPI; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy (Experimental): Patients with rectal cancer will receive short-course radiotherapy and neoadjuvant chemotherapy plus immunotherapy.
  68Ga-FAPI-04 and 18F-FDG PET will be performed at baseline and after short-course radiotherapy and 2 cycles of neoadjuvant chemotherapy plus immunotherapy. The two imaging intervals will be completed two days apart.
  Interventions: Drug: 68Ga-FAPI-04; Drug: 18F-FDG

INTERVENTIONS:
Drug: 68Ga-FAPI-04 — A fibroblast activation protein (FAP) -targeted PET imaging agent
  Other Names: 68Ga-FAPI
Drug: 18F-FDG — A general glucose metabolism imaging agent
  Other Names: 18F-fluorodeoxyglucose

SUMMARY:
This study is a prospective monocentric study aimed to explore the value of 68Ga-FAPI-04 PET imaging in early response evaluation of rectal cancer patients treated with immunotherapy. Patients with histopathologically confirmed diagnosis of rectal cancer will be recruited and undergo 68Ga-FAPI-04 and 18F-FDG PET imaging before treatment and after short-course radiotherapy and two cycles of neoadjuvant chemotherapy plus immunotherapy. The two imaging intervals will be completed two days apart. The efficacy of 68Ga-FAPI-04 in early response evaluation will be compared with the general imaging agent 18F-FDG. The general information, clinical data, mpMRI data, 68Ga-FAPI-04 and 18F-FDG PET imaging results and other imaging data of the patients will be collected. The histopathology of the biopsy or surgical specimen after 2 cycles of therapy and follow-up data will be taken as evaluation references. This study plans to set the sample size as 20 cases

DETAILED DESCRIPTION:
The response patterns of immune checkpoint inhibitors (ICIs) in solid tumors are diverse and complicated. Pseudoprogression, progression and even hyperprogression can occur. The main mechanism of pseudoprogression is the infiltration of immune cells into the tumor lesion, causing blurred tumor margins and even an increase in the volume of the entire tumor lesion (secondary delayed response). For pseudoprogression, irRC, irRECIST, iRECIST and other immune-related solid tumor efficacy evaluation criteria based on anatomical images are not enough to confirm, and the inflammation caused by T cell infiltration also shows strong uptake of 18F-FDG. The existing criteria for the response evaluation in solid tumors cannot early identify progression or pseudoprogression.

Fibroblast activation protein (FAP) is highly specifically expressed on the membrane surface of carcinoma-associated fibroblast (CAF). FAP-positive CAFs exist in a variety of solid tumors including rectal cancer and are mainly involved in the formation of tumor stroma. However, FAP is rarely expressed in normal tissues. Therefore, 68Ga-FAPI-04 PET, a FAP-targeted imaging modality, can be used to differentiate tumors and normal tissues and has been widely used in clinical studies. Its sensitivity and specificity outperformed 18F-FDG PET. Studies have shown that tumors with high FAP expression are associated with poor response immunotherapy. Although FAP-targeted imaging has been widely used in predicting the response to immune checkpoint inhibitors, it has rarely been reported in rectal cancer.

This study is a prospective monocentric study aimed to explore the value of 68Ga-FAPI-04 PET imaging in the early response evaluation of rectal cancer patients treated with immunotherapy. Patients with histopathologically confirmed diagnosis of rectal cancer will be recruited and undergo 68Ga-FAPI-04 and 18F-FDG PET imaging before treatment and after short-course radiotherapy and two cycles of neoadjuvant chemotherapy plus immunotherapy. The two imaging intervals will be completed two days apart. The efficacy of 68Ga-FAPI-04 in early response evaluation will be compared with the general imaging agent 18F-FDG.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed T3-4N0M0 or T1-4N+M0 (according to the 8th edition of the International Union Against Cancer TNM staging system) rectal adenocarcinoma and treatment naïve;
* No severe hematologic, cardiac, pulmonary, hepatic, or renal functional abnormalities or immunodeficiency diseases;
* An Eastern Cooperative Oncology Group Performance Status of 0-1;
* Patients who agree to undergo 68Ga-FAPI-04 and 18F-FDG PET imaging.

Exclusion Criteria:

* Any experiences of anti-programmed death ligand 1 (PD-L1) or anti-PD-1 antibody treatment;
* A history of pelvic radiation;
* The presence of autoimmune disease;
* Hypersensitive to any monoclonal antibodies;
* History of interstitial lung disease;
* Active and uncontrolled infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
68Ga-FAPI-04 PET analysis | Baseline and 21-28 days after 2 cycles of neoadjuvant chemotherapy plus immunotherapy (each cycle is 21-28 days)
  PET parameter (SUVmax in g/ml, MTV in cm3, TLG in g/ml×cm3, etc.) changes between both scans will be measured.
18F-FDG PET analysis | Baseline and 21-28 days after 2 cycles of neoadjuvant chemotherapy plus immunotherapy (each cycle is 21-28 days)
  PET parameter (SUVmax in g/ml, MTV in cm3, TLG in g/ml×cm3, etc.) changes between both scans will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- China, Hubei Province, Wuhan, Hubei, China